CLINICAL TRIAL: NCT03246399
Title: A Phase 1, Open-label Study of the Safety, Tolerability, and Pharmacokinetics of SM04690 Injectable Suspension Following Single Intradiscal Injection in Subjects With Degenerative Disc Disease
Brief Title: A Study of the Safety, Tolerability, and Pharmacokinetics of SM04690 Injectable Suspension Following Single Intradiscal Injection in Subjects With Degenerative Disc Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped due to business reasons, following full enrollment of the first dose cohort.
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SM04690-DDD-01
Record Dates: First submitted 2017-06-29; First posted 2017-08-11 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Degenerative Disc Disease
Keywords: SM04690; Wnt pathway; Samumed
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — lorecivivint

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.03mg SM04690 (Experimental): 0.03mg SM04690 per 0.5 mL intradiscal injection (single injection at Day 1)
  Interventions: Drug: SM04690
- 0.07mg SM04690 (Experimental): 0.07mg SM04690 per 0.5 mL intradiscal injection (single injection at Day 1)
  Interventions: Drug: SM04690
- 0.15mg SM04690 (Experimental): 0.15mg SM04690 per 0.5 mL intradiscal injection (single injection at Day 1)
  Interventions: Drug: SM04690

INTERVENTIONS:
Drug: SM04690 — suspension formulation of SM04690, delivered via intradiscal injection (single injection)

SUMMARY:
SM04690-DDD-01 is a Phase 1, open-label, dose escalation study. SM04690 Injectable Suspension will be administered via a single intradiscal injection to subjects with degenerative disc disease (DDD) under fluoroscopic guidance. Groups of 6 subjects will be enrolled in successive cohorts. Subjects will participate in a 6 month follow-up period. Clinic visits will be Screening, Treatment Visit Day 1, and Follow-up Visit Days 2, 15, 28, 60, 90, 135, and 180.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative disease in a maximum of two and a minimum of one lumbar disc (L4/L5 or L5/S1)
* Persistent low back pain due to DDD for at least 3 months prior to study start
* Full understanding of the requirements of the study and willingness to comply with all study visits and assessments
* Subjects must have read and understood the informed consent form, and must have signed it prior to any study-related procedure being performed

Exclusion Criteria:

* Women who are pregnant, lactating, or have a positive pregnancy result at study start
* Women of child bearing potential who are sexually active and are not willing to use a highly effective method of birth control during the study period
* Males who are sexually active and have a partner who is capable of becoming pregnant, neither of whom have had surgery to become sterilized or whom are not using a highly effective method of birth control
* Body mass index (BMI) > 35
* Previous participation in a Samumed clinical trial investigating SM04690
* History of compression fractures and/or osteoporosis
* Any herniation in the lumbar spine as identified by MRI
* Congenital or acquired diseases leading to spine deformations
* History of hypersensitivity or allergies to any ingredient of the study medication
* Participation in a clinical research trial that included the receipt of an investigational product or any experimental therapeutic procedure, or an observational research trial related to DDD within 8 weeks prior to any study injection, or planned participation in any such trial; the last date of participation in the trial, not the last date of receipt of investigational product, must be at least 8 weeks prior to study start
* Poor peripheral venous access
* Any contraindications to MRI according to MRI guidelines
* History of malignancy; however, subjects with prior history of in situ cancer or basal or squamous cell skin cancer, completely cured, are eligible.
* Any diagnosed psychiatric condition that includes, but is not limited to, a history of mania, bipolar disorder, psychotic disorder, schizophrenia, schizoaffective disorder, major depressive disorder, or generalized anxiety disorder
* Prior surgical procedures (e.g., discectomy, intradiscal electrothermal therapy, intradiscal radiofrequency, artificial disc replacement, and interbody fusion) on the lumbar spine
* Any planned or elective surgery during the study period
* Any known active infections, including hepatitis B or hepatitis C infection, and/or infections that may compromise the immune system such as human immunodeficiency virus (HIV)
* Current or prior history of any spinal infection (i.e., discitis, septic arthritis, or epidural abscess)
* Any lumbar intradiscal injection procedure (e.g., injection of corticosteroids, methylene blue, dextrose, etc.), myelograms, discography, and/or lumbar epidural or transforaminal injections with corticosteroids or nerve-blocking anesthetics (e.g, lidocaine, bupivacaine) within 3 months prior to study start
* Any electrotherapy (i.e., transcutaneous electrical nerve stimulation [TENS] unit) or acupuncture for DDD within 4 weeks prior to study medication injection
* History of or current/pending disability claim, workers' compensation, or litigation(s) related to back pain/injury
* Subjects who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at any investigative site, or are directly affiliated with the study at any investigative site
* Subjects employed by Samumed, LLC, or any of its affiliates or development partners (that is, an employee, temporary contract worker, or designee) responsible for the conduct of the study, or who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of said employees responsible for the conduct of the study

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: treatment emergent adverse events (TEAEs) | Day 180
  Evaluate the safety and tolerability of SM04690 Injectable Suspension as measured by TEAEs during the entire treatment and observation period
Safety and tolerability: change from baseline in electrocardiogram (ECG) parameters | Baseline and Day 180
  Evaluate the safety and tolerability of SM04690 Injectable Suspension as measured by change from baseline in ECG parameters
Safety and tolerability: change from baseline in physical examination | Baseline and Day 180
  Evaluate the safety and tolerability of SM04690 Injectable Suspension as measured by change from baseline in physical examination (number of subjects with clinically significant change in physical examination)
Safety and tolerability: change from baseline in clinical laboratory tests | Baseline and Day 180
  Evaluate the safety and tolerability of SM04690 Injectable Suspension as measured by change from baseline in clinical laboratory tests (number of subjects with clinically significant changes in laboratory test parameters)
Safety and tolerability: change from baseline in vital signs | Baseline and Day 180
  Evaluate the safety and tolerability of SM04690 Injectable Suspension as measured by change from baseline in vital signs (number of subjects with clinically significant changes in vital signs)
Incidence of dose-limiting toxicities (DLTs) | Day 180
  Evaluate incidence and severity of DLTs in each cohort
Pharmacokinetics (PK) of SM04690: Cmax | Day 1
  Maximum plasma concentration (Cmax) estimate for a single intradiscal injection of SM04690 Injectable Suspension
PK of SM04690: tmax | Day 1
  Time to Cmax estimate for a single intradiscal injection of SM04690 Injectable Suspension
PK of SM04690: AUC | Day 1
  Area under the plasma-concentration time curve (AUC) estimate for a single intradiscal injection of SM04690 Injectable Suspension
PK of SM04690: half-life | Day 1
  Plasma terminal phase half-life estimate for a single intradiscal injection of SM04690 Injectable Suspension

SECONDARY OUTCOMES:
Change in spine bone mineral density | Baseline and Day 180
  Evaluate change from baseline spine bone mineral density as measured by dual-energy x-ray absorptiometry (DXA)
Change in hip bone mineral density | Baseline and Day 180
  Evaluate change from baseline hip bone mineral density as measured by DXA

OTHER OUTCOMES:
Change in lumbar back pain | Baseline and Day 180
  Evaluate change from baseline lumbar back pain using the Visual Analog Scale (VAS)
Change in disability | Baseline and Day 180
  Evaluate change from baseline disability as measured by Oswestry disability index (ODI)
Change in disease activity by physician assessment | Baseline and Day 180
  Evaluate change from baseline disease activity using Physician Global Assessment (PGA)
Change in treated intervertebral discs | Baseline and Day 180
  Evaluate change from baseline in treated intervertebral discs by modified Pfirrmann grade using Magnetic Resonance Imaging (MRI)
Change in disc space height | Baseline and Day 180
  Evaluate change from baseline in disc space height by radiograph

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (4):
- United States (4):
  - Research Site, San Diego, California
  - Research Site, Charleston, South Carolina
  - Research Site, Tyler, Texas
  - Research Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No